CLINICAL TRIAL: NCT06780969
Title: Breastfeeding: A Sustainable Choice to Reduce Carbon Footprint
Brief Title: A Sustainable Choice to Reduce Carbon Footprint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Leyla Kaya, Assoc. Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 06.09.2023/118
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; Carbon footprint; Sustainability; Nutrition; Environmental impact
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Women selected for the experimental group will receive 4 sessions of Green Mother Training.
  The programme, which includes breastfeeding, bonding and carbon footprint training, is delivered 4 times by researchers.
  The training content has been prepared by the researchers by scanning the literature. The training will be delivered using posters.
  Interventions: Behavioral: Green Mother Training
- Control (No Intervention): Women in the control group receive routine care at the same hospital's polyclinics.

INTERVENTIONS:
Behavioral: Green Mother Training — Poster education
  Arms: Experimental

SUMMARY:
This study aimed to evaluate the impact of carbon footprint education on breastfeeding practices among pregnant women.

DETAILED DESCRIPTION:
This study aimed to evaluate the impact of carbon footprint education on breastfeeding practices among pregnant women.

In the sample size calculation performed using G*Power 3.1.9.7 (Faul et al., 2007) software, the effect size value determined for the relationship between awareness levels regarding sustainable and healthy nutrition behaviors and reducing ecological footprint was determined as Cohen's r=0.470. Statistical power analysis was performed under A Priori: Compute required sample size (Correlation: Bivariate normal model), 95% power (1-β) and α=0.05 and in the light of these parameters, it was concluded that a sample size of at least 53 participants was required for the study in question. In case of data loss, it was envisaged to increase the sample by 20% as a result of statistical consultancy. Accordingly, it was planned to conduct the study with a total of n=64 people, n=32 in the intervention group and n=32 in the control group.

It was carried out with the participation of two groups. The carbon footprint education group received 4 education sessions of 60 minutes each. The control group received routine hospital care during this period, but no other intervention was made.

Data for the study were collected by the researcher using face-to-face interviews, a personal information form with demographic questions, and the measurement tools used in the study. The training was completed 4 weeks later. After the training, the measurement tools were used for the woman's postpartum period.

Participants were given an explanation of the carbon footprint education and told how, for how long, and where the education would take place. The carbon footprint education programme was completed by the participants in a specific way (nutrition, breastfeeding, environmental awareness) for each session. The education was delivered using a poster.

The carbon footprint education was given in 4 sessions in this way. The measurement tools were given to the participants again on the 1st day, 1st month, 3rd month and 6th month after birth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 24 weeks gestation
* Must be between 18 and 35 years of age.
* Women must provide informed consent to participate in the study, indicating their willingness to participate in the educational intervention and assessments.
* Attend educational sessions

Exclusion Criteria:

* Women with significant medical conditions that may affect breastfeeding or nutrition (e.g. serious mental illness, chronic disease) will be excluded.
* Multiple pregnancies
* Previous GREEN MOTHER training
* Substance abuse
* Women considered to be at high risk of non-compliance with the study protocol (e.g. those with unstable living conditions).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Famale
Enrollment: 100 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Scale Breast-feeding Self-efficacy Scale | 1st day after birth, 3rd month after birth, 6th month after birth
  Breastfeeding Self-Efficacy Scale: This is a 33-item scale developed by Dennis (1999). It consists of two sub-dimensions to determine mothers' breastfeeding skills, beliefs and behaviours regarding breastfeeding. The validity and reliability study of the Turkish form of the scale was conducted by Ekşioğlu and Çeber (2011). Breastfeeding self-efficacy was assessed using a five-point Likert scale: (1) I never trust myself, (2) I do not trust myself very much, (3) I trust myself sometimes, (4) I trust myself often, (5) I always trust myself. As the total score on the scale increases, so does breastfeeding self-efficacy. The lowest score is 33 and the highest is 165.
Ecological Footprint Awareness Scale | Participants immediately after group assignment, 6 months after the birth
  The Ecological Footprint Awareness Scale consists of six sub-dimensions: energy, legal, recycling, transport, water use and food. The scale categories are obtained by summing the subscales and scoring them as strongly disagree=1, disagree=2, undecided=3, agree=4 and strongly agree=5. The Cronbach's alpha value was found to be 0.960.
Behaviors Scale Towards Sustainable Nutrition | Participants immediately after group assignment, 6 months after the birth
  The developed scale consists of 29 items and 4 sub-dimensions with a five-point Likert scale. It includes the sub-dimensions of food preference, reducing food waste, eating seasonally and locally, and buying food. The scale is rated as 'never', 'rarely', 'sometimes', 'often' and 'always'. All items are scored from 1 to 5, starting with 'never'. All items in the scale are positive. The lowest score that can be obtained from the scale is 29 and the highest score is 145. Sub-dimension scores are obtained by dividing the sum of the scores given by individuals to the questions in the sub-dimension by the number of questions in the sub-dimension. Higher total and sub-dimension scores indicate that the individual has more sustainable dietary behaviours.
Depression Anxiety and Stress scales-21 (DASS-21) | Participants immediately after group assignment, 1st day after delivery, 3rd month after delivery, 6th month after delivery
  his 21-item scale consists of three dimensions, namely anxiety, depression, and stress. Items are measured on a 4-point Likert-type scale ranging from 0 (Never) to 3 (Always). A higher sum score indicates more severe symptoms of depression, anxiety, and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Keles, PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No